CLINICAL TRIAL: NCT04177537
Title: Efficacy of SAM Sport as an Addon to Traditional Therapy in Treating Sports-related Injuries
Brief Title: Real-World Experience of Athletes Treated With SAM
Status: Completed | Type: Observational
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AL-01
Record Dates: First submitted 2019-11-11; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Pain, Chronic; Pain, Acute; Sport Injury; Soft Tissue Injuries; Arm Injury; Back Pain; Tendon Injuries; Muscle Injury
Keywords: low-intensity ultrasound; continuous ultrasound; long-duration ultrasound; athletic training; clinical trial; soft tissue; pain; Musculoskeletal tissue; ZetrOZ System LLC
MeSH Terms: conditions — Chronic Pain; Acute Pain; Soft Tissue Injuries; Arm Injuries; Back Pain; Tendon Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Pre-Low Intensity Continuous Ultrasound Treatment: Retrospective analysis of pain alleviation, range of motion and ability to return to work with traditional therapies selected from one rehabilitation facility
- Post-Low Intensity Continuous Ultrasound Treatment: Retrospective analysis of pain alleviation, range of motion and ability to return to work after treatment with low-intensity continuous ultrasound (LICUS) in conjunction with traditional therapies selected from one rehabilitation facility
  Interventions: Device: Low Intensity Continuous Ultrasound

INTERVENTIONS:
Device: Low Intensity Continuous Ultrasound — 3MHz, 0.132W/cm2, 1.3W for 4 hours day delivered by an acoustic device provided by Zetroz Systems LLC
  Groups: Post-Low Intensity Continuous Ultrasound Treatment

SUMMARY:
Low-intensity continuous ultrasound (LICUS) is an FDA-approved bio regenerative technology, applied with a wearable device (SAM, Zetroz Systems LLC) for daily use. The treatment provides long-duration ultrasound for approximately four hours. This report included a retrospective convenience sample of 6 athletes from one sports medicine and rehabilitation facility. The objective of this report is to examine the real-world outcome data on symptoms improvement and return to function using Sam. It was hypothesized that LICUS stimulation, in conjunction with traditional therapies, will accelerate the healing process of musculoskeletal tissue leading to a reduction in pain, increase functionality, and a higher probability of returning to work and sports-related activities. The sample included athletes with sports-related musculoskeletal injuries. Demographics, injury history, treatment history, and clinical outcomes data were retrospectively collected for athletes who were treated with SAM in conjunction with traditional therapies. Clinical results showed a benefit from the treatment with a decrease in pain (100%), and 3 out of 6 athletes were able to return to work or sports (50%). Overall the study shows that Sam accelerates the healing of soft tissue leading to a decrease in both acute and chronic pain.

DETAILED DESCRIPTION:
The cohort of 6 male athletes (n=6) ages ranged from 18 to 54 years of age, with an average age of 33.5 years with musculoskeletal injuries, which showed little or no improvement with traditional therapies selected from one rehabilitation facility. The group included 3 amateur athletes and 3 professional athletes participated in baseball (2) and golf (1). No healthy athlete was selected, considering the study of nature.

Demographic, injury history, treatment history, and clinical outcomes data of the patients were collected. The patients were asked about the effectiveness of traditional therapies such as physical therapy, manual therapy, a combination of rest, ice, compression, and elevation (RICE). The athletes with sports-related musculoskeletal related injuries, including arm, upper leg, back, quadriceps, knees, foot/ankles, were treated with low-intensity continuous ultrasound (SAM®, ZetrOZ Sysmtem LLC device) in conjunction with traditional therapies. At that point, data were recorded, and patients were advised to use LICUS in conjunction with conventional therapies. The athletes were asked about the effectiveness of LICUS treatment as an add-on to traditional therapies. Furthermore, .the effectiveness of the treatment was assessed by patient response to pain relief, range of motion, and ability to going back to the sport.

The LICUS was delivered by easy to use wearable LICUS device (SAM®, ZetrOZ Systems, LLC, Trumbull, CT) consisting of two transducers powered by an external battery pack was used to deliver at 3MHz, 0.132W/cm2, 1.3W for 4 hours. The athletes were trained to use the device using ultrasound coupling gel on the injured area. It was ensured that all the athletes knew how to use the device properly. The device is easy to use with three buttons setup: an on/off button (middle), a time, and on/off lock buttons on the sides.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with musculoskeletal injuries with limited improvement under traditional therapies

Exclusion Criteria:

* Healthy Athletes

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Athletes with sport-related musculoskeletal injuries.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NRS) (0-10) | variable (1 - 8 weeks)
  Change in pain severity over the time of treatment, 0 being lowest, and 10 being the worst pain. A total of 6 athletes were examined through questionnaires. in which they were asked about the change of pain on the NRS scale. No adverse effects were reported throughout the study.

OTHER OUTCOMES:
Return to Work on the scale of number of week | variable (1 - 8 weeks)
  Athletes reported response to a questionnaire, implying the return to sporting activity, the lowest number of weeks means quicker recovery and a higher number of weeks meant the lowest recovery

CONTACTS AND LOCATIONS:
Overall Officials: David O Draper, EdD, Study Chair — Brigham Young University

REFERENCES:
- [Result] Heckman JD, Ryaby JP, McCabe J, Frey JJ, Kilcoyne RF. Acceleration of tibial fracture-healing by non-invasive, low-intensity pulsed ultrasound. J Bone Joint Surg Am. 1994 Jan;76(1):26-34. doi: 10.2106/00004623-199401000-00004. PMID 8288661
- [Result] Zhang N, Chow SK, Leung KS, Cheung WH. Ultrasound as a stimulus for musculoskeletal disorders. J Orthop Translat. 2017 Apr 5;9:52-59. doi: 10.1016/j.jot.2017.03.004. eCollection 2017 Apr. PMID 29662799
- [Result] Best TM, Wilk KE, Moorman CT, Draper DO. Low Intensity Ultrasound for Promoting Soft Tissue Healing: A Systematic Review of the Literature and Medical Technology. Intern Med Rev (Wash D C). 2016 Dec;2(11):271. doi: 10.18103/imr.v2i11.271. PMID 30198009
- [Result] Langer MD, Lewis GK Jr. Sustained Acoustic Medicine: A Novel Long Duration Approach to Biomodulation Utilizing Low Intensity Therapeutic Ultrasound. Proc SPIE Int Soc Opt Eng. 2015 May;9467:94670I. doi: 10.1117/12.2178213. PMID 30078928
- [Result] Lewis GK Jr, Langer MD, Henderson CR Jr, Ortiz R. Design and evaluation of a wearable self-applied therapeutic ultrasound device for chronic myofascial pain. Ultrasound Med Biol. 2013 Aug;39(8):1429-39. doi: 10.1016/j.ultrasmedbio.2013.03.007. Epub 2013 Jun 4. PMID 23743101
- [Result] Rigby JH, Taggart RM, Stratton KL, Lewis GK Jr, Draper DO. Intramuscular Heating Characteristics of Multihour Low-Intensity Therapeutic Ultrasound. J Athl Train. 2015 Nov;50(11):1158-64. doi: 10.4085/1062-6050-50.11.03. Epub 2015 Oct 28. PMID 26509683
- [Result] Enwemeka CS, Rodriguez O, Mendosa S. The biomechanical effects of low-intensity ultrasound on healing tendons. Ultrasound Med Biol. 1990;16(8):801-7. doi: 10.1016/0301-5629(90)90044-d. PMID 2095010
- [Result] Nolte PA, van der Krans A, Patka P, Janssen IM, Ryaby JP, Albers GH. Low-intensity pulsed ultrasound in the treatment of nonunions. J Trauma. 2001 Oct;51(4):693-702; discussion 702-3. doi: 10.1097/00005373-200110000-00012. PMID 11586161
- [Result] Jia XL, Chen WZ, Zhou K, Wang ZB. Effects of low-intensity pulsed ultrasound in repairing injured articular cartilage. Chin J Traumatol. 2005 Jun;8(3):175-8. PMID 15896276
- [Result] D'Vaz AP, Ostor AJ, Speed CA, Jenner JR, Bradley M, Prevost AT, Hazleman BL. Pulsed low-intensity ultrasound therapy for chronic lateral epicondylitis: a randomized controlled trial. Rheumatology (Oxford). 2006 May;45(5):566-70. doi: 10.1093/rheumatology/kei210. Epub 2005 Nov 22. PMID 16303817
- [Result] Khanna A, Nelmes RT, Gougoulias N, Maffulli N, Gray J. The effects of LIPUS on soft-tissue healing: a review of literature. Br Med Bull. 2009;89:169-82. doi: 10.1093/bmb/ldn040. Epub 2008 Nov 16. PMID 19011263
- [Result] Fu SC, Hung LK, Shum WT, Lee YW, Chan LS, Ho G, Chan KM. In vivo low-intensity pulsed ultrasound (LIPUS) following tendon injury promotes repair during granulation but suppresses decorin and biglycan expression during remodeling. J Orthop Sports Phys Ther. 2010 Jul;40(7):422-9. doi: 10.2519/jospt.2010.3254. PMID 20479531
- [Result] Nagata K, Nakamura T, Fujihara S, Tanaka E. Ultrasound modulates the inflammatory response and promotes muscle regeneration in injured muscles. Ann Biomed Eng. 2013 Jun;41(6):1095-105. doi: 10.1007/s10439-013-0757-y. Epub 2013 Feb 6. PMID 23386031
- [Result] Draper DO, Ricard MD. Rate of Temperature Decay in Human Muscle Following 3 MHz Ultrasound: The Stretching Window Revealed. J Athl Train. 1995 Oct;30(4):304-7. PMID 16558352
- [Result] Alexander LD, Gilman DR, Brown DR, Brown JL, Houghton PE. Exposure to low amounts of ultrasound energy does not improve soft tissue shoulder pathology: a systematic review. Phys Ther. 2010 Jan;90(1):14-25. doi: 10.2522/ptj.20080272. Epub 2009 Nov 12. PMID 19910457
- [Result] Best TM, Moore B, Jarit P, Moorman CT, Lewis GK. Sustained acoustic medicine: wearable, long duration ultrasonic therapy for the treatment of tendinopathy. Phys Sportsmed. 2015 Nov;43(4):366-74. doi: 10.1080/00913847.2015.1095617. Epub 2015 Oct 15. PMID 26468991
- See also: Conference Proceedings Volume 1113, Issue 1, p.403-407 — https://ui.adsabs.harvard.edu/abs/2009AIPC.1113..403L/abstract
- See also: Conference Proceedings Volume publication date 15 August 2004 — https://www.annualreviews.org/doi/abs/10.1146/annurev.bioeng.6.040803.140126